CLINICAL TRIAL: NCT04040049
Title: A Phase 1/2, Baseline-controlled, Non-randomized, Open-label, Single-ascending Dose Study of a Novel Adeno-associated Viral Vector (FLT190) in Patients With Fabry Disease
Brief Title: A Fabry Disease Gene Therapy Study
Acronym: MARVEL1
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Freeline has decided to pause development of FLT190 in Fabry disease to focus its resources on advancing FLT201.
Sponsor: Spur Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FLT190-01
Record Dates: First submitted 2019-07-26; First posted 2019-07-31 (Actual); Last update posted 2023-06-05 (Actual); Status verified 2023-04

CONDITIONS: Fabry Disease; Lysosomal Storage Diseases
Keywords: Gene Therapy
MeSH Terms: conditions — Fabry Disease; Lysosomal Storage Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- FLT190 (Experimental): FLT190 is a recombinant adeno- associated viral (AAV) vector. Administered by a single intravenous infusion.
  Interventions: Genetic: FLT190

INTERVENTIONS:
Genetic: FLT190 — Gene Therapy product.

SUMMARY:
This is a multinational, open-label study to assess the safety and efficacy of FLT190 in up to 15 adult male participants with classical Fabry disease.

DETAILED DESCRIPTION:
Patients who provide consent to participate in this study will be screened for eligibility.

Eligible patients will attend the study site on the day prior to infusion (Day -1) for a baseline visit. On Day 0, FLT190 will be administered as a single dose, slow intravenous infusion. Following FLT190 treatment the patient will be discharged from the investigational site and will continue to be monitored at outpatient visits for a period of approximately 9 months; following which, the patient will enter a period of long-term follow-up conducted under a separate protocol.

The study will be conducted in 2 parts;

Part 1: Enrolment of previously treated patients (Dose escalation)

Part 2: Enrolment of previously untreated patients (Dose expansion).

ELIGIBILITY:
Inclusion Criteria:

1. Adult males, ≥ 18 years of age with classic Fabry disease.
2. Confirmed diagnosis of classic Fabry Disease
3. Decreased plasma alpha galactosidase (αGLA) activity at screening.
4. One or more of the characteristic features of classic Fabry disease.
5. Estimated glomerular filtration rate (eGFR) ≥60mL/min/1.73m2 at screening.
6. <500 mg/g Urine Protein to Creatinine Ratio (UPCR) in a spot urine sample OR < 1g/24 hours of urinary protein (24hour urine analysis), at
7. Able to give full informed consent and able to comply with all requirements of the trial including the 5-year long term follow-up.
8. Willingness to practice barrier contraception whilst vector shedding via semen is present.
9. Lack of AAV neutralizing antibodies within 6 weeks prior to dosing.
10. For inclusion in Part 1, subjects must have received either a licensed ERT or PCT for at least 12 months prior to dosing. For inclusion in Part 2, subjects must never have been previously dosed with Enzyme Replacement Therapy (ER) or Pharmacological Chaperone Therapy (PCT).
11. Willingness to avoid strenuous exercise during first 3 months after dosing.

Exclusion Criteria:

1. Non-classical Fabry disease.
2. Prior hypersensitivity or intolerance to ERT
3. Prior lack of response to ERT.
4. Subjects with a history of chronic kidney disease for a minimum of 3 months.
5. Subjects with severe myocardial fibrosis.
6. Use of investigational therapy for Fabry disease within 60 days before enrolment. In addition, participation in any other clinical trial of an investigational medicinal product (IMP), and/or receiving any other IMP during the course of the study
7. Evidence of liver dysfunction as demonstrated by elevated blood levels during screening.
8. Platelet count < 100 xE9L.
9. Subjects receiving warfarin or other anticoagulants or subjects with a clinically significant bleeding disorder.

10 - 12. Either history of, or a positive serology test at screening for hepatitis B surface antigen (HBsAg), hepatitis B core antibody (HBcAb), hepatitis C antibody (HCAb) and human immunodeficiency virus (HIV) or a negative test at screening for anti-varicella zoster virus (VZV) IgG or hepatitis surface antibody (HBsAb).

13. Subjects with a history of or a positive screening test for tuberculosis. 14. Subjects who have received a live attenuated vaccination within 12 weeks prior to screening or intend to receive such a vaccine within the course of the study.

15. Uncontrolled glaucoma, diabetes mellitus, or hypertension. 16. History of any malignancy requiring treatment. 17. History or detection of significant arrhythmia during screening. 18. Subjects with uncontrolled cardiac failure, unstable chest pain, or heart attack deemed significant in the past 6 months.

19. History of acute myocarditis or presence of acute myocarditis during screening.

20. Prior treatment with any gene therapy medicinal product. 21. Known or suspected intolerance to gadolinium, tacrolimus and other macrolides, steroids, local anesthetics used for skin or renal biopsies, or any non-investigational medicinal products (NIMPs) or their excipients.

22. Subjects with contraindications to MRI. Including subjects with ferromagnetic metallic implants, including pacing and defibrillator devices, nerve stimulators and cochlear implants.

23. Subjects who have had a renal transplant. 24. Cytomegalovirus immunoglobulin positive subjects who are CMV polymerase chain reaction (PCR) positive at screening.

25-26.History of physical or psychiatric illness that could affect the subject's ability to participate or a history of substance abuse including alcohol abuse.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2019-07-08 (Actual); Primary Completion 2023-05-02 (Actual); Study Completion 2023-05-02 (Actual)

PRIMARY OUTCOMES:
Frequency of treatment-emergent adverse events (AEs) | From screening to 12 weeks post infusion
  To investigate the safety of systemic administration of FLT190.

CONTACTS AND LOCATIONS:
Locations (13):
- United States (4):
  - Kaiser Permanente, Los Angeles, California
  - Columbia University, New York, New York
  - UPMC Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Lysosomal and Rare Disorders Research and Treatment Center, Fairfax, Virginia
- Medical University of Vienna, Vienna, Austria
- Metabolics and Genetics in Calgary (MAGIC Clinic), Calgary, Toronto, Canada
- Germany (3):
  - Charité - Universitätsmedizin Berlin, Berlin
  - UKEA University Hospital Hamburg, Hamburg
  - University of Würzburg, Würzburg
- Universita Federico II di Napoli, Napoli, Italy
- Haukeland University Hospital, Bergen, Norway
- United Kingdom (2):
  - Royal Free Hospital, London
  - Salford Royal NHS Foundation Trust, Salford

REFERENCES:
- [Derived] Jeyakumar JM, Kia A, Tam LCS, McIntosh J, Spiewak J, Mills K, Heywood W, Chisari E, Castaldo N, Verhoef D, Hosseini P, Kalcheva P, Cocita C, Miranda CJ, Canavese M, Khinder J, Rosales C, Hughes D, Sheridan R, Corbau R, Nathwani A. Preclinical evaluation of FLT190, a liver-directed AAV gene therapy for Fabry disease. Gene Ther. 2023 Jun;30(6):487-502. doi: 10.1038/s41434-022-00381-y. Epub 2023 Jan 11. PMID 36631545